CLINICAL TRIAL: NCT02008617
Title: Analgesic Benefits of Genicular Nerve Blocks of the Posterior Knee for Patients Undergoing Anterior Cruciate Ligament (ACL) Reconstruction
Brief Title: Analgesic Benefits of Genicular Nerve Blocks of the Posterior Knee for Patients Undergoing ACL Reconstruction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated due to lack of subject recruitment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Rohit Rahangdale, Assistant Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU00085894; STU00085894
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: Anterior cruciate ligament reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Drug (Active Comparator): Ultrasound guided posterior genicular nerve infiltration with 30mL of Bupivicaine 0.20% with epinephrine 1:300,000 (Study Drug)
  Interventions: Drug: Bupivacaine
- Preservative free normal saline (Sham Comparator): Ultrasound guided posterior genicular nerve infiltration posterior knee with 30mL of preservative free normal saline
  Interventions: Drug: Preservative free normal saline

INTERVENTIONS:
Drug: Bupivacaine — 30mL of Bupivicaine 0.20% with epinephrine 1:300,000
  Other Names: Marcaine
  Arms: Study Drug
Drug: Preservative free normal saline — Ultrasound guided posterior genicular nerve infiltration posterior knee with 30mL of preservative free normal saline
  Other Names: 0.9% sodium chloride
  Arms: Preservative free normal saline

SUMMARY:
Outpatients scheduled to have ACL surgery typically receive a femoral nerve block to provide analgesia for the front of the knee. Postoperatively, these patients will often report pain in the back of the knee. Local anesthetic infiltration of the posterior aspect of the knee results in blockade of the genicular nerves of the posterior knee. These nerves originate off of the tibial and common peroneal nerves and their blockade will result in improved posterior knee pain relief and may decrease narcotic consumption compared to patients who receive the same infiltration with normal saline.

DETAILED DESCRIPTION:
Femoral nerve blocks are commonly used to provide postoperative analgesia for ACL surgery. The limitation of these blocks is the incomplete analgesia they provide of the knee joint subjecting the patient to posterior knee pain. As a result, some of these patients receive rescue sciatic blocks in the postoperative care unit to cover posterior knee pain. The sciatic block provides excellent analgesia for the posterior knee; however its blockade invariably affects other territories of the sciatic nerve such as the lower leg and foot. For ACL surgery, the loss of sensation and/or motor strength to this area is unnecessary and may make ambulation more difficult. The ability to ambulate with minimal assistance may be more important for a patient undergoing an outpatient surgery when compared to an inpatient surgery.

At the posterior knee, the sciatic nerve branches off into the tibial and common peroneal nerves which give rise to sensory fibers that innervate the posterior knee. We propose targeting these terminal fibers in the popliteal fossa by infiltrating local anesthetic between the distal femoral shaft and popliteal artery thereby providing posterior knee analgesia without affecting the lower leg.This application of this block has not been studied in patients having ACL surgery. A single interim analysis is scheduled after the data for 50 cases are available.

ELIGIBILITY:
Inclusion Criteria:

1. patients who are presenting for ACL reconstruction
2. candidates for peripheral nerve blocks patients
3. ASA 1-3

Exclusion Criteria:

1. Patient refusal
2. ASA Classification of 4 or higher
3. Pre-existing neuropathy in the femoral or sciatic distribution
4. Coagulopathy
5. Infection at the site
6. Non-English speaking or non-reading patients
7. Chronic opioid use (>3months)
8. Pregnancy
9. Any other contra-indication to regional anesthesia
10. Failed femoral nerve block
11. Sciatic nerve block placed due to severe pain not managed by intravenous and oral agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Rahangdale, M.D., Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Drug: Ultrasound guided posterior genicular nerve infiltration with 30mL of Bupivicaine 0.20% with epinephrine 1:300,000
  Bupivacaine: 30mL of Bupivicaine 0.20% with epinephrine 1:300,000
Period: Overall Study
Arm/Group | Study Drug | Preservative Free Normal Saline
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Drug | Preservative Free Normal Saline | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25 [24 to 32] | 29 [23 to 38] | 27 [23 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption
Description: Opioid consumption (mg morphine equivalents)
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalents
Arm/Group | Study Drug | Preservative Free Normal Saline
Number analyzed (Participants) | 8 | 10
mg morphine equivalents | 50 [40 to 70] | 70 [50 to 80]
Statistical Analysis 1: Comparison: Study Drug vs Preservative Free Normal Saline; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Pain Score
Description: Numeric Rating Scale (NRS) (NRS pain scores; 0 = no pain,10 = excruciating pain) in the back of the knee recorded every 4 hours up to 24hrs following surgery. Pain Bruden scale ranges from 0 (no pain) to 240 (extreme pain). For example, pain burden of 120 is equivalent to a NRS score of 5 out of 10.
Time Frame: Pain Burden at 24hrs
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Study Drug | Preservative Free Normal Saline
Number analyzed (Participants) | 8 | 10
units on a scale
  Pain Score at Rest | 102 [58 to 160] | 135 [112 to 146]
  Pain Score during plantar flexion | 115 [50 to 182] | 128 [96 to 144]
Statistical Analysis 1: Comparison: Study Drug vs Preservative Free Normal Saline; At Rest; Test type: Superiority or Other; p = 0.86, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Study Drug vs Preservative Free Normal Saline; Plantar Flexion; Test type: Superiority or Other; p = 0.89, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction with pain control scale ranges from 0 (no satisfaction) to 10 (very satisfied).
Time Frame: 24hr
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Study Drug | Preservative Free Normal Saline
Number analyzed (Participants) | 8 | 10
units on a scale | 8 [7 to 8] | 8 [6 to 10]
Statistical Analysis 1: Comparison: Study Drug vs Preservative Free Normal Saline; Test type: Superiority or Other; p = 0.78, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Quality of Recovery (QoR15)
Description: Quality of recovery (QoR15) is a questionnaire that asks 15 questions regarding how the participant has felt in the last 24 hours. Each question is followed by an 11-point numerical rating scale (0 = "none of the time" to 10 = "all of the time"; maximum score 150). The higher the QoR15 total score, the worse the quality of recovery reported.
Time Frame: 24hrs
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Study Drug | Preservative Free Normal Saline
Number analyzed (Participants) | 8 | 10
units on a scale | 96 [84 to 110] | 102 [80 to 114]
Statistical Analysis 1: Comparison: Study Drug vs Preservative Free Normal Saline; Test type: Superiority or Other; p = 0.82, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 24hr following surgery.
Arm/Group | Study Drug | Preservative Free Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes